CLINICAL TRIAL: NCT06772012
Title: Effectiveness of Low-Level Laser Therapy (LLLT) Versus Orofacial Physical Therapy for Temporomandibular Dysfunction. a Randomized Controlled Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahria University (Other)
Responsible Party: Principal Investigator, Seyyada Tahniat Ali, physiotherapist, Bahria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU92-MSRSW-F22-085
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Temporomandibular Dysfunction
Keywords: temporomandibular dysfunction
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-Level Laser Therapy (LLLT) (Experimental): Intervention Protocol:
  * Frequency: LLLT was administered 3 times per week.
  * Duration: Each session lasted approximately 15-20 minutes.
  * Total Duration: The therapy was provided for a total of 6 weeks.(50)
  Interventions: Other: Low-Level Laser Therapy (LLLT)
- Orofacial Physical Therapy (Active Comparator): Intervention Protocol:
  * Frequency: Orofacial physical therapy sessions were conducted 3 times per week.
  * Duration: Each session lasted around 30-40 minutes.
  * Total Duration: The therapy was provided for a total of 6 weeks.
  * Components:
    * Manual Therapy: Included techniques such as joint mobilization, soft tissue manipulation, and muscle stretching.
    * Therapeutic Exercises: Focused on strengthening, coordination, and improving mobility of the masticatory muscles.
    * Postural Training: Addressed poor posture and cervical muscle spasm.(50)
  Interventions: Other: Orofacial Physical Therapy

INTERVENTIONS:
Other: Low-Level Laser Therapy (LLLT) — * Frequency: LLLT was administered 3 times per week.
  * Duration: Each session lasted approximately 15-20 minutes.
  * Total Duration: The therapy was provided for a total of 6 weeks.(50)
  Arms: Low-Level Laser Therapy (LLLT)
Other: Orofacial Physical Therapy — * Frequency: Orofacial physical therapy sessions were conducted 3 times per week.
  * Duration: Each session lasted around 30-40 minutes.
  * Total Duration: The therapy was provided for a total of 6 weeks.
  * Components:
    * Manual Therapy: Included techniques such as joint mobilization, soft tissue manipulation, and muscle stretching.
    * Therapeutic Exercises: Focused on strengthening, coordination, and improving mobility of the masticatory muscles.
    * Postural Training: Addressed poor posture and cervical muscle spasm.(50)
  Arms: Orofacial Physical Therapy

SUMMARY:
This study will investigate if Low-Level Laser Therapy (LLLT) is more effective than Orofacial Physical Therapy for treating Temporomandibular Dysfunction. By conducting a randomized controlled trial, it aims to fill gaps in current knowledge, improve TMD treatment options, and enhance patient outcomes.

DETAILED DESCRIPTION:
In the last 30 years, many nonsurgical therapies have been suggested for the treatment of temporomandibular disorders (TMD), including physical therapy, pharmacologic therapy, occlusal splints, occlusal adjustment, acupuncture, and low-level laser therapy (LLLT). (1) The main objective of all these treatment modalities is to reduce symptom intensity, thereby improving the function of the masticatory system and adjacent structures.(2) Signs and symptoms of TMD are present in 86% of the population, being more frequent among women, also related to dental occlusion and emotional stress. Are considered signs: limited mouth opening, joint sounds and deviation of the mandible to one side during opening and closing, muscle spasm, pain reflex, impaired joint motion, crepitus, headache and hearing disorders. Otologic symptoms are represented by decreased hearing, vertigo and tinnitus, which can be related to the ontogenetic and anatomical relationship between the middle ear and masticatory structures.(3) Among nonsurgical treatments, LLLT has increased in interest in the last few years, probably due to its ease of use in combination with reports of positive effects on pain alleviation. (4) LLLT is a non-thermal type of light, which causes internal changes in cells and tissues, leading to different types of metabolic activations. (5) These include stimulation of the cellular respiratory chain and increase in vascularization and fibroblast formation which have been suggested to play an important role in the analgesic effect of LLLT. Despite the fact that there is no universally accepted theory to explain the mechanism of either "laser analgesia" or "laser bio stimulation,"(6) LLLT can be expected to promote some anti-inflammatory effect and pain relief in painful and dysfunctional joints and muscles.(7) The most clinically used LLLT include the helium-neon laser (632 nm He-Ne) and infrared laser, as diode-gallium-arsenide (904 nm Ga-As) or gallium-aluminium-arsenide (830 nm Ga-Al-As). The mechanism of pain relief via mid-laser therapy is not clearly understood and several theories have been suggested. One theory considers the analgesic effect to be a consequence of the reduction of levels of prostaglandin E2 (PGE2 ), which is one of the most important proinflammatory mediators. This theory is based on in vivo and in vitro findings of a reduction of PGE2 both in cultures of ligament cells and in the joint capsule of animals after laser exposure. The PGE2 reduction probably derives from the inhibition made by laser radiation of cyclooxygenase-2 (COX-2), the enzyme involved in the synthesis of PGE.(8, 9) Another theory takes into account the effect of laser therapy on neuronal cells: The effect involves the possible selective inhibition of nociceptive signals16 and the microcirculation regulation; this action could interrupt the origin and development of pain and thus could provide analgesic effects.17,18 The magnitude of the laser effect seems to depend on the wavelength and dosage of the laser light.11 It has been reported that reduction of PGE2 could be observed within a range of dose between 0.4 and 19 J and within a range of power density between 5 and 21.2 mW/cm2 . (10)

Temporomandibular disorders (TMDs) are probably the most common cause of pain of non-dental origin in the maxillofacial area. The category of TMDs embraces a number of clinical problems related to masticator muscles, temporomandibular joint (TMJ) and associated structures, or both. (11) Such disorders are characterised by pain, joint sounds, and restricted mandibular movement. The incidence of TMD ranges from 40 to 75 % in general populations and approximately 65 % of affected patients experience associated pain. This great number of patients is treated using different modalities, depending on the aetiology of signs and symptoms. Conservative, rather than aggressive and irreversible, treatment is preferred to relieve symptoms, diminish pain, and re-establish function. (12, 13) As the aetiology of TMD is multifactorial, available treatments are extensive and diverse, including the use of occlusal splints, low-level laser therapy (LLLT), and transcutaneous electrical nerve stimulation, among many others. Given that better therapeutic results (i.e. pain relief ) are obtained with the combined use of modalities, several recent studies have examined the use of LLLT to reduce TMD pain and promote bio augmentation effects. (14) The LLT has demonstrated an ability to assist in the symptomatic treatment of pain, providing a considerable degree of comfort to the patient after application. The great advantage of laser applications in the treatment of TMD is that it is a non-invasive therapy, with low cost, and currently has being widely used in dental practice, reducing the demand related to the surgery or the use of drugs to treat relief pain and tissue regeneration.(15) The application of laser therapy in TMD patients has demonstrated an ability to relieve pain in few minutes after application, promoting well-being significant. However, LLT is an adjuvant treatment in pain relief by its analgesic action, which allows the patient's return to daily chores, providing comfort and better quality of life.(16) The G1 group was randomly divided into 7 therapeutic groups in which the therapy was carried out for 10 days: magneto stimulation (T1), magnetoledotherapy (T2), magnetolaserotherapy (T3), manual therapy- positional release and therapeutic exercises (T4), manual therapy - massage and therapeutic exercises (T5), manual therapy - PIR and therapeutic exercises (T6), self therapy - therapeutic exercises (T7).G2 was given LLLT. (17) Most people can open their mouth 35 to 55 millimeters (1.4 to 2.2 inches), which is about the width of 3 fingers (see Figure 2). Figure 2. Normal width of an open mouth Your jaw is made up of a pair of bones that form the framework of your mouth and teeth.(18)

This study will investigate if Low-Level Laser Therapy (LLLT) is more effective than Orofacial Physical Therapy for treating Temporomandibular Dysfunction. By conducting a randomized controlled trial, it aims to fill gaps in current knowledge, improve TMD treatment options, and enhance patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 1) limited mouth opening or function(49) 2) presence of pain in masticatory muscles and/or TMJs(49) 3) muscular disturbance (49) 4) arthralgia(49)

Exclusion Criteria:

* 1) major systemic disorders (49) 2) who received analgesic or anti-depressants over the last 2 weeks(49) 3) had any bony abnormalities of the jaws (49) 4) psychological illness (49) 5) pregnant and feeding women (49)

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
jaw range of motion | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Bahria University, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petrucci A, Sgolastra F, Gatto R, Mattei A, Monaco A. Effectiveness of low-level laser therapy in temporomandibular disorders: a systematic review and meta-analysis. J Orofac Pain. 2011 Fall;25(4):298-307. PMID 22247925